CLINICAL TRIAL: NCT01066884
Title: A Study of First or Second Line Treatment With Tarceva (Erlotinib) in Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML20569
Record Dates: First submitted 2010-02-04; First posted 2010-02-10 (Estimated); Last update posted 2016-08-24 (Estimated); Status verified 2016-08

CONDITIONS: Non-Squamous Non-Small Cell Lung Cancer
MeSH Terms: interventions — Erlotinib Hydrochloride

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: erlotinib [Tarceva]

INTERVENTIONS:
Drug: erlotinib [Tarceva] — 150mg po daily

SUMMARY:
This single arm study will assess the safety and efficacy of Tarceva monotherapy in patients with advanced non-small cell lung cancer. Patients will receive Tarceva 150mg p.o. daily. The anticipated time on study treatment is until disease progression, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >= 18 years of age;
* inoperable, locally advanced, recurrent or metastatic (Stage IIIB/IV) non-small cell lung cancer;
* ECOG performance status of 0-3;
* previously untreated, or failed on one prior course of standard systemic chemotherapy and/or radiotherapy.

Exclusion Criteria:

* prior systemic anti-tumor therapy with HER1/EGFR inhibitors;
* unstable systemic disease;
* any other malignancies within 5 years (except for adequately treated cancer in situ of the cervix, or basal or squamous cell skin cancer;
* any significant ophthalmologic abnormality.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2009-04; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | Length of patient on study (length of time of patient on study determined by investigator)

SECONDARY OUTCOMES:
Best Response Rate per investigator assessment | Length of patient on study (length of time of patient on study determined by investigator)
Time to Progression (TTP) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first
Overall survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (2):
- Russia (2):
  - Balashikha
  - Krasnoyarsk